CLINICAL TRIAL: NCT00033826
Title: The Role of Adipose Tissue in Vitamin D Metabolism
Brief Title: Role of Fat Tissue in Vitamin D Metabolism
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Miriam Blum, MD, HNRC at Tufts
Other Study IDs: K23AR047869 (NIH); K23AR047869 (NIH); NIAMS-070
Record Dates: First submitted 2002-04-10; First posted 2002-04-11 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Vitamin D; Adipose Tissue
Keywords: Vitamin D; Adipose tissue; Metabolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Vitamin D is a fat soluble vitamin that has important effects on calcium (including absorption of calcium from the diet) and bone metabolism. Vitamin D is known to be stored in fat tissue, and it is also present in the circulation. The purpose of this study is to investigate the relationship between levels of vitamin D in fat tissue and in blood.

DETAILED DESCRIPTION:
Although vitamin D is known to be stored in fat tissue, researchers are not sure about the role that fat tissue plays in vitamin D metabolism. This study will help develop the methodology necessary to further investigate the role of fat tissue in vitamin D metabolism and will assess the relationship between levels of vitamin D in fat tissue and in blood. 50 subjects who are referred for gastric bypass surgery will be enrolled in this study. Subjects will complete questionnaires about their medical history, travel history and food intake. Prior to or during surgery, subjects will be asked to provide a blood sample for selected chemistries related to vitamin D metabolism. During gastric bypass surgery, the surgeon will collect small pieces of fat tissue from the fat under the skin and within the abdomen by surgical biopsy. These samples will be used to refine the methodology for determining the levels of vitamin D in blood and fat tissue and for comparing levels of vitamin D in various tissues.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients referred for gastric bypass surgery

Exclusion Criteria:

* Patients must not be taking bile acid-sequestering medications or anti-seizure medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from Obesity Clinic
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2002-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Blum, MD, Principal Investigator — Jean Mayer USDA Human Nutrition Center on Aging at Tufts University
Locations (1):
- Tufts-New England Medical Center, Boston, Massachusetts, United States